CLINICAL TRIAL: NCT03010072
Title: The Effect of Phosphate Lowering Using Sucroferric Oxyhydroxide (PA21) on Calcification Propensity of Serum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prim. Priv. Doz. Dr. Daniel Cejka (Other)
Collaborators: Vifor Fresenius Medical Care Renal Pharma (Industry)
Responsible Party: Sponsor-Investigator, Prim. Priv. Doz. Dr. Daniel Cejka, Prim. Priv. Doz. Dr., Elisabethinen Hospital
Organization: Elisabethinen Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PA21-T50-CKD5D
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Endstage Renal Disease
MeSH Terms: interventions — sucroferric oxyhydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose sucroferric oxyhydroxide (Active Comparator): Low dose 250 mg sucroferric oxyhydroxide (PA21) per day (1x 250mg tablets/day) for 14 days.
  Interventions: Drug: low-dose sucroferric oxyhydroxide
- high-dose sucroferric oxyhydroxide (Active Comparator): Uniform dose 2000 mg of sucroferric oxyhydroxide (PA21) per day (4x 500mg tablets/day) for 14 days
  Interventions: Drug: high-dose sucroferric oxyhydroxide

INTERVENTIONS:
Drug: low-dose sucroferric oxyhydroxide — 250 mg suroferric oxyhydroxide
  Other Names: suroferric oxyhydroxide tablets; Velphoro
  Arms: low-dose sucroferric oxyhydroxide
Drug: high-dose sucroferric oxyhydroxide — 2000 mg suroferric oxyhydroxide
  Other Names: suroferric oxyhydroxide tablets; Velphoro
  Arms: high-dose sucroferric oxyhydroxide

SUMMARY:
This is a single-center, prospective, open-label, controlled, randomized, cross-over study in 34 prevalent end-stage renal disease patients on chronic hemodialysis treatment with hyperphosphatemia.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio to either receive low-dose (250mg/d) PA-21 followed by high-dose (2000mg/d) PA-21 (sequence A-B) or to receive high-dose PA21 followed by low-dose PA21 (sequence B-A) with washout-phases in between. An open label design with a sub-therapeutic dose of PA21 as control treatment was chosen because creating a convincing placebo for PA21 is not feasible.

The study will start with two study visits on the 2nd and 3rd dialysis session of the week , where dialysis patients are still treated with standard of care to establish baseline values (duration: 0.5 weeks). Next will be an initial run-in wash-out phase, where all phosphate binders taken by the patient as standard of care treatment will be discontinued and no phosphate binders will be introduced. Consequently, there will be a PA21 treatment (high dose/low dose) phase, followed by a wash-out phase, followed by another PA21 treatment (high dose/low dose) phase, followed by a final wash-out phase. Each study phase, including wash-out phases as well as low-dose and high-dose treatment phases will be 14 days of duration. Patients will be followed up to 10.5 weeks after randomization until the last study visit of the final wash-out phase.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent patients (≥ 3 months on dialysis) treated with thrice weekly hemodialysis (HD) or hemodiafiltration (HDF)
* Hyperphosphatemia (serum phosphate > upper limit of normal within the last 3 months) or current phosphate binder use
* No use or constant dose of vitamin D and/or calcimimetics for ≥2 weeks

Exclusion Criteria:

* Allergy to sucroferric oxyhydroxide (PA21), to other ingredients of Velphoro or to any iron-medication
* Current or history of calciphylaxis (calcific uremic arteriolopathy - CUA)
* parathormone >800 pg/ml
* Parathyreoidektomie planned or expected
* Significant GI or hepatic disorders
* Hypercalcemia (total serum calcium >2.6 mmol/l) at screening
* Antacids containing aluminum, calcium, magnesium or bicarbonate
* Oral iron treatments/supplements
* Pregnant and nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Propensity of serum for calcification - H1 | 10.5 weeks
  The primary outcome is change in the mean T50- Test values between different study phases (wash-out/treatment/control).

SECONDARY OUTCOMES:
Change in Serum Phosphate | 10.5 weeks
  The secondary outcome is the Change of mean Serum Phosphate Levels between different study visits

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cejka, Dr., Principal Investigator — Sponsor/PI
Locations (1):
- Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No